CLINICAL TRIAL: NCT01374282
Title: Post Marketing Surveillance Study of Cuprimine (MK-0172-001)
Brief Title: Post Marketing Surveillance Study of Cuprimine
Status: No longer available | Type: Expanded Access
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0172-001
Record Dates: First submitted 2011-06-14; First posted 2011-06-15 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Penicillamine

INTERVENTIONS:
Drug: Cuprimine (penicillamine) — Dosage determined by the physician based on indication for treatment

SUMMARY:
Cuprimine (penicillamine) was made available in the Philippines by the Sponsor under a Compassionate Special Permit issued by the Bureau of Food and Drugs. Physicians were able to request the drug for their patients from the Sponsor. A Clinical Study Report form was completed for each purchase of Cuprimine.

ELIGIBILITY:
Inclusion Criteria:

- None

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult